CLINICAL TRIAL: NCT05584202
Title: A Phase 2, Two-Part Study (Open-Label [Part 1] Followed by Observer-Blind/Randomized [Part 2]) to Evaluate the Safety, Tolerability, Reactogenicity, and Effectiveness of mRNA-1273.214 SARS-CoV-2 Vaccine in Participants Aged 12 Weeks to < 6 Months
Brief Title: Study to Evaluate the Safety, Reactogenicity, and Effectiveness of mRNA-1273.214 SARS-CoV-2 (COVID-19) Vaccine in Infants
Acronym: BabyCOVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated because data from the dose finding part of the trial did not support further evaluation of effectiveness of mRNA-1273. There were no safety concerns.
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1273-P206
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; mRNA-1273.214 vaccine; mRNA-1273.214; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID 19; COVID 19 Vaccine; Moderna; Bivalent omicron vaccine; Omicron vaccine
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19 | interventions — mRNA-1273.214 COVID-19 vaccine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Part 1: sequential Part 2: parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1: open-label Part 2: observer-blinded, randomized, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: mRNA-1273.214 Dose A (Experimental): Participants will receive 2 doses of mRNA-1273.214 Dose A by intramuscular (IM) injection approximately 8 weeks apart (Day 1 and Day 57).
  Interventions: Biological: mRNA-1273.214
- Part 1: mRNA-1273.214 Dose B (Experimental): Participants will receive 2 doses of mRNA-1273.214 Dose B by IM injection approximately 8 weeks apart (Day 1 and Day 57).
  Interventions: Biological: mRNA-1273.214
- Part 2: mRNA-1273.214 (Experimental): Participants will receive 2 doses of mRNA-1273.214 by IM injection approximately 8 weeks apart (Day 1 and Day 57).
  Interventions: Biological: mRNA-1273.214
- Part 2: Placebo (Placebo Comparator): Participants will receive 2 doses of placebo by IM injection approximately 8 weeks apart (Day 1 and Day 57).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: mRNA-1273.214 — Sterile liquid for injection
  Arms: Part 1: mRNA-1273.214 Dose A; Part 1: mRNA-1273.214 Dose B; Part 2: mRNA-1273.214
Other: Placebo — 0.9% sodium chloride
  Other Names: normal saline
  Arms: Part 2: Placebo

SUMMARY:
The study evaluated the safety, tolerability, reactogenicity, and effectiveness of mRNA-1273.214 severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine in infants aged 12 weeks to < 6 months.

DETAILED DESCRIPTION:
The purpose of this pediatric study was to confirm safety and effectiveness of mRNA-1273.214 in infants between 12 weeks to < 6 months of age by comparing the immune response of infants in this study to adults (>18 years of age) enrolled in the mRNA-1273-P301 study [NCT04470427]).

The study was planned to be conducted in 2 parts. Part 1 was open-label and evaluated 2 dose levels. The dose level selected from Part 1 was planned to be further evaluated in Part 2. However, data from the dose finding part of the trial (Part 1) did not support further evaluation of effectiveness of mRNA-1273 and accordingly, Part 2 of the study was not conducted and the trial was terminated. There were no safety concerns.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is male or female, between 2 and <6 months of age at the time of consent (Screening Visit), who is in good general health, in the opinion of the investigator, based on review of medical history and screening physical examination.

  1. Participant must be at least 12 weeks completed age and must not have completed 6 months at the time of administration of first dose.
  2. If the participant has a chronic, stable disease, they may be eligible to enroll in Part 2, but ineligible for Part 1. The chronic condition (for example, gastroesophageal reflux disease) should be stable, per investigator assessment, so that the participant can be considered eligible for inclusion in Part 2.
* Participant was born at ≥37 weeks gestation (Part 1) or ≥34 weeks gestation (Part 2), with a minimum birth weight of 2.5 kilograms (kg), without fetal growth restriction, and the participant's height and weight are both at or above the second percentile for age according to the Centers for Disease Control and Prevention/World Health Organization Child Growth Standard at the Screening Visit.
* In the investigator's opinion, the parent(s)/legally authorized representative(s) understand and are willing and physically able to comply with protocol-mandated follow-up, including all procedures, and provide written informed consent.

Key Exclusion Criteria:

* Participant has a known history of SARS-CoV-2 infection within 2 weeks prior to administration of study drug or has a known close contact in the past 2 weeks to someone diagnosed with SARS-CoV-2 infection or coronavirus disease 2019 (COVID-19). Participants may be rescreened after 14 days provided that they remain asymptomatic.
* Participant is acutely ill or febrile 72 hours prior to or at the Screening Visit. Fever is defined as a body temperature ≥38.0°Celcius/≥100.4°Farenheit. Participants who meet this criterion may have visits rescheduled within the relevant study visit windows. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator.
* Participant has previously been administered an investigational or approved CoV (for example, SARS-CoV-2, SARS-CoV, Middle East respiratory syndrome [MERS]-CoV) vaccine.
* Participant has undergone treatment with investigational or approved agents for prophylaxis against COVID-19 (for example, receipt of SARS-CoV-2 monoclonal antibodies) within 90 days prior to enrollment.
* Participant has a known hypersensitivity to a component of the vaccine or its excipients. Hypersensitivity includes, but is not limited to, anaphylaxis or immediate allergic reaction of any severity to any of the components of messenger ribonucleic acid (mRNA) COVID-19 vaccines (including polyethylene glycol or immediate allergic reaction of any severity to polysorbate).
* Participant has a medical, psychiatric, or occupational condition, that, according to the investigator's judgment, may pose additional risk as a result of participation, interfere with safety assessments, or interfere with interpretation of results.
* Participant has a history of diagnosis or condition that, in the judgment of the investigator, may affect study endpoint assessment or compromise participant safety.
* Participant has received the following:

  1. Any routine vaccination with inactivated or live vaccine(s) within 14 days prior to first or second vaccination or plans to receive such a vaccine within 14 days of any study vaccination.
  2. Systemic immunosuppressants or immune-modifying drugs (including maternal use during pregnancy or lactation) for >14 days in total within 6 months prior to the day of enrollment (for corticosteroids, ≥ 1 milligrams (mg)/kg/day or, if participant weighs >10 kg: ≥10 mg/day prednisone equivalent). Participants may have visits rescheduled for enrollment if they no longer meet this criterion within the Screening Visit window. Inhaled, nasal, and topical steroids are allowed.
  3. Intravenous or subcutaneous blood products (red blood cells, platelets, immunoglobulins) within 3 months prior to enrollment.
* Participant has participated in an interventional clinical study within 28 days prior to the Screening Visit or plans to do so while participating in this study, or maternal participation in an interventional clinical study during pregnancy.

Note: Other inclusion and exclusion criteria may apply.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Trinity Clinical Research, LLC - Bessemer, Bessemer, Alabama
  - UAB Pediatrics, Birmingham, Alabama
  - Eclipse Clinical Research, Tucson, Arizona
  - Madera Family Medical Group, Madera, California
  - SeraCollection Research Services LLC, Montebello, California
  - Center For Clinical Trials LLC, Paramount, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Meridian Clinical Research (Washington) - PPDS, Washington D.C., District of Columbia
  - PAS Research, Clearwater, Florida
  - Prohealth Research Center, Doral, Florida
  - University of Florida Jackonsville, Jacksonville, Florida
  - Kissimmee Clinical Research, Kissimmee, Florida
  - Acevedo Clinical Research, Miami, Florida
  - D&H National Research Centers, Miami, Florida
  - Suncoast Research Associates LLC - ERN - PPDS, Miami, Florida
  - Excellence Medical and Research LLC, Miami Gardens, Florida
  - KM International Research Operation - Saint Cloud, Saint Cloud, Florida
  - PAS Research, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Medical Research Partners- Ammon, Ammon, Idaho
  - MedPharmics - Platinum - PPDS, Covington, Louisiana
  - MedPharmics - Platinum - PPDS, Lafayette, Louisiana
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Clinical Research Institute, Inc, Minneapolis, Minnesota
  - Be Well Clinical Studies, Lincoln, Nebraska
  - Child Health Care Associates, East Syracuse, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Velocity Clinical Research (Hastings - Nebraska) - PPDS, Wilmington, North Carolina
  - UPMC University Center, Pittsburgh, Pennsylvania
  - Coastal Pediatric Research, Charleston, South Carolina
  - South Texas Clinical Research - Corpus Christi, Corpus Christi, Texas
  - Cedar Health Research - Dedicated Research Facility, Dallas, Texas
  - DM Clinical Research - Kool Kids Pediatrics - ERN - PPDS, Houston, Texas
  - Advances In Health Inc, Pearland, Texas
  - Victoria Clinical Research Group, Port Lavaca, Texas
  - Tanner Clinic, Layton, Utah
  - Wee Care Pediatrics, Syracuse, Utah
  - PI-Coor Clinical Research LLC, Burke, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants eligible for enrollment in Part 1 of this study included male and female infants aged 12 weeks to <6 months at the time of administration of first dose who were in good general health.
Groups:
- mRNA-1273.214 5 μg: Participants received at least 1 of the 2 doses of mRNA-1273.214 5 micrograms (μg) by intramuscular (IM) injection approximately 8 weeks apart (Day 1 and Day 57).
- mRNA-1273.214 10 μg: Participants received at least 1 of the 2 doses of mRNA-1273.214 10 μg by IM injection approximately 8 weeks apart (Day 1 and Day 57).
Period: Overall Study
Arm/Group | mRNA-1273.214 5 μg | mRNA-1273.214 10 μg
Started | 50 | 18
Received First Injection | 50 | 18
Received Second Injection | 49 | 15
Safety Set (Safety Set included participants who received at least 1 dose of study drug.) | 50 | 18
Solicited Safety Set First Injection (Solicited Safety Set (First Injection) included participants who received the first injection of study drug and contributed any solicited adverse reaction (AR) data.) | 50 | 18
Solicited Safety Set Second Injection (Solicited Safety Set (Second Injection) included participants who received the second injection of study drug and contributed any solicited AR data.) | 49 | 15
Per-Protocol Immunogenicity Set (PPIS) (PPIS included participants who received the planned doses of investigational product per schedule, complied with immunogenicity testing schedule, had Baseline (Day 1) and Day 85 antibody assessments, and had no major protocol deviations that impacted key or critical data.) | 37 | 11
Completed | 45 | 14
Not Completed | 5 | 4
Not completed — Withdrawal of Consent | 3 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Groups:
- mRNA-1273.214 5 μg: Participants received at least 1 of 2 doses of mRNA-1273.214 5 μg by IM injection approximately 8 weeks apart (Day 1 and Day 57).
- mRNA-1273.214 10 μg: Participants received at least 1 of 2 doses of mRNA-1273.214 10 μg by IM injection approximately 8 weeks apart (Day 1 and Day 57).
- Total: Total of all reporting groups
Arm/Group | mRNA-1273.214 5 μg | mRNA-1273.214 10 μg | Total
Number analyzed (Participants) | 50 | 18 | 68
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 50 | 18 | 68
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 4 | 30
  Male | 24 | 14 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 6 | 18
  Not Hispanic or Latino | 38 | 12 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 35 | 9 | 44
  Race: Black or African American | 13 | 5 | 18
  Race: Asian | 1 | 0 | 1
  Race: Multiracial | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs) After First Injection
Description: Solicited ARs (local and systemic) were collected in an electronic diary (eDiary). Local ARs included injection site pain/tenderness, injection site erythema (redness), injection site swelling/induration (hardness), and groin or underarm swelling or tenderness ipsilateral to the side of injection. Systemic ARs included fever, irritability/crying, sleepiness, and loss of appetite. Solicited AR severity was graded according to a modified version (relevant to age 12 weeks to <6 months) of the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials. ARs graded 1-4 are presented. Lower scores indicated lower severity, and higher scores indicated greater severity. A summary of serious adverse events (SAEs) and nonserious adverse events (AEs) (Safety Set), regardless of causality, is located in the AE section.
Time Frame: Day 1 up to 7 days after first vaccination (up to Day 8)
Population: Solicited Safety Set (First Injection) included participants who received the first injection of study drug and contributed any solicited AR data.
Measure: Count of Participants; unit: Participants
Groups:
- mRNA-1273.214 5 μg First Injection (Solicited Safety Set): Participants received first injection of mRNA-1273.214 5 μg.
- mRNA-1273.214 10 μg First Injection (Solicited Safety Set): Participants received first injection of mRNA-1273.214 10 μg.
Arm/Group | mRNA-1273.214 5 μg First Injection (Solicited Safety Set) | mRNA-1273.214 10 μg First Injection (Solicited Safety Set)
Number analyzed (Participants) | 50 | 18
Participants
  Grade 1 | 23 | 7
  Grade 2 | 8 | 3
  Grade 3 | 1 | 0
  Grade 4 | 0 | 0
  Any solicited ARs (Grade 1-4) | 32 | 10

2. Primary Outcome: Number of Participants With Solicited Local and Systemic ARs After Second Injection
Description: Solicited ARs (local and systemic) were collected in eDiary. Local ARs included injection site pain/tenderness, injection site erythema (redness), injection site swelling/induration (hardness), and groin or underarm swelling or tenderness ipsilateral to the side of injection. Systemic ARs included fever, irritability/crying, sleepiness, and loss of appetite. Solicited AR severity was graded according to a modified version (relevant to age 12 weeks to <6 months) of the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials. ARs graded 1-4 are presented. Lower scores indicated lower severity, and higher scores indicated greater severity. A summary of SAEs and nonserious AEs (Safety Set), regardless of causality, is located in the AE section.
Time Frame: Day 57 up to 7 days after second vaccination (up to Day 64)
Population: Solicited Safety Set (Second Injection) included participants who received the second injection of study drug and contributed any solicited AR data.
Measure: Count of Participants; unit: Participants
Groups:
- mRNA-1273.214 5 μg Second Injection (Solicited Safety Set): Participants received second injection of mRNA-1273.214 5 μg.
- mRNA-1273.214 10 μg Second Injection (Solicited Safety Set): Participants received second injection of mRNA-1273.214 10 μg.
Arm/Group | mRNA-1273.214 5 μg Second Injection (Solicited Safety Set) | mRNA-1273.214 10 μg Second Injection (Solicited Safety Set)
Number analyzed (Participants) | 49 | 15
Participants
  Grade 1 | 18 | 6
  Grade 2 | 7 | 2
  Grade 3 | 1 | 0
  Grade 4 | 0 | 0
  Any solicited ARs (Grade 1-4) | 26 | 8

3. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs) After Any Injection
Description: An unsolicited AE was any AE reported by the participant that was not specified as a solicited AR in the protocol or was specified as a solicited AR but started outside the protocol-defined period for reporting solicited ARs (onset after Day 7 of dosing). An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result or other safety assessment, including one that worsened from baseline and was considered clinically significant by the Investigator was recorded as an AE. A summary of SAEs and nonserious AEs (Safety Set), regardless of causality, is located in the AE section. COVID-19/SARS-CoV-2 infections were considered clinical events and not AEs.
Time Frame: Day 1 up to 28 days after any vaccination (up to Day 85)
Population: Safety Set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- mRNA-1273.214 5 μg (Safety Set): Participants received at least 1 of 2 doses of mRNA-1273.214 5 μg by IM injection approximately 8 weeks apart (Day 1 and Day 57).
- mRNA-1273.214 10 μg (Safety Set): Participants received at least 1 of 2 doses of mRNA-1273.214 10 μg by IM injection approximately 8 weeks apart (Day 1 and Day 57).
Arm/Group | mRNA-1273.214 5 μg (Safety Set) | mRNA-1273.214 10 μg (Safety Set)
Number analyzed (Participants) | 50 | 18
Participants | 24 | 8

4. Primary Outcome: Number of Participants With SAEs, AEs of Special Interest (AESIs), Medically Attended AEs (MAAEs), and AEs Leading to Study or Treatment Discontinuation
Description: SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs were identified based upon medical concepts that may be related to COVID-19 or were of interest in COVID-19 vaccine safety surveillance. MAAE was an AE that led to an unscheduled visit to a healthcare practitioner, included visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up, and visits to healthcare practitioners external to the study site [for example, urgent care, primary care physician]). A summary of SAEs and nonserious AEs (Safety Set), regardless of causality, is located in the AE section. COVID-19/SARS-CoV-2 infections were considered clinical events and not AEs.
Time Frame: Day 1 up to Day 422
Population: Safety Set included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1273.214 5 μg (Safety Set) | mRNA-1273.214 10 μg (Safety Set)
Number analyzed (Participants) | 50 | 18
Participants
  SAEs | 1 | 1
  AESIs | 1 | 0
  MAAEs | 39 | 16
  AEs Leading to Study or Treatment Discontinuation | 0 | 1

5. Secondary Outcome: Geometric Mean Concentration (GMC) of Serum Pseudovirus Neutralizing Antibod (nAb) Titers Against SARS-CoV-2 Omicron BA.1 Variant (B.1.1.529) After Second Dose of mRNA-1273.214
Description: Pseudovirus nAb were measured using pseudovirus neutralization assay (PsVNA). Antibody values reported as below the lower limit of quantification (LLOQ) were replaced by 0.5*LLOQ. Values greater than the upper limit of quantification (ULOQ) were replaced by the ULOQ if actual values were not available. VAC122 nAb against the SARS-CoV-2 B.1.1.529 variant (LLOQ: 8 arbitrary unit (AU)/milliliter (mL), ULOQ: 24503 AU/mL).
Time Frame: Baseline and 28 days after second dose (Day 85)
Population: PPIS: participants who received the planned doses of investigational product per schedule, complied with immunogenicity testing schedule, had Baseline (Day 1) and Day 85 antibody assessments, and had no major protocol deviations that impacted key or critical data.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Groups:
- mRNA-1273.214 5 μg (PPIS): Participants received the planned doses of mRNA-1273.214 5 μg per schedule, complied with immunogenicity testing schedule, had Baseline (Day 1) and Day 85 antibody assessments, and had no major protocol deviations that impacted key or critical data.
- mRNA-1273.214 10 μg (PPIS): Participants received the planned doses of mRNA-1273.214 10 μg per schedule, complied with immunogenicity testing schedule, had Baseline (Day 1) and Day 85 antibody assessments, and had no major protocol deviations that impacted key or critical data.
Arm/Group | mRNA-1273.214 5 μg (PPIS) | mRNA-1273.214 10 μg (PPIS)
Number analyzed (Participants) | 37 | 11
AU/mL
  Baseline | 64.9 [42.3 to 99.6] | 84.2 [42.8 to 165.5]
  Day 85 | 163.0 [91.0 to 292.2] | 228.6 [97.0 to 538.9]

6. Secondary Outcome: GMC of Serum Pseudovirus nAb Titers Against SARS-CoV-2 Original Strain (D614G) After Second Dose of mRNA-1273.214
Description: Pseudovirus nAb were measured using PsVNA assay. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. VAC62 Neutralizing Antibody against D614G (LLOQ: 10 AU/mL, ULOQ: 111433 AU/mL).
Time Frame: Baseline and 28 days after second dose (Day 85)
Population: PPIS: participants who received the planned doses of investigational product per schedule, complied with immunogenicity testing schedule, had Baseline (Day 1) and Day 85 antibody assessments, and had no major protocol deviations that impacted key or critical data. Number analyzed = participants evaluable for the specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | mRNA-1273.214 5 μg (PPIS) | mRNA-1273.214 10 μg (PPIS)
Number analyzed (Participants) | 37 | 11
AU/mL
  Baseline | 236.4 [150.8 to 370.6] | 203.6 [76.6 to 540.9]
  Day 85: number analyzed (Participants) | 36 | 11
  Day 85 | 178.1 [133.3 to 237.9] | 96.0 [72.2 to 127.6]

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 422
Description: Safety Set included participants who received at least 1 dose of study drug.
Groups:
- mRNA-1273.214 5 ug: Participants received at least 1 of 2 doses of mRNA-1273.214 5 μg by IM injection approximately 8 weeks apart (Day 1 and Day 57).
- mRNA-1273.214 10 ug: Participants received at least 1 of 2 doses of mRNA-1273.214 10 μg by IM injection approximately 8 weeks apart (Day 1 and Day 57).
Arm/Group | mRNA-1273.214 5 ug | mRNA-1273.214 10 ug
All-Cause Mortality (participants affected / at risk) | 0/50 | 1/18
Serious Adverse Events (participants affected / at risk) | 1/50 | 1/18
Other Adverse Events (participants affected / at risk) | 40/50 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mRNA-1273.214 5 ug (N=50) | mRNA-1273.214 10 ug (N=18)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) — Cardiac arrest resulting from drowning in the 10 ug group.
Drowning (General disorders) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) — Hypoxic-ischaemic encephalopathy resulting from drowning in the 10 ug group.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mRNA-1273.214 5 ug (N=50) | mRNA-1273.214 10 ug (N=18)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 6 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 2 (4)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 6 (7) | 1 (1)
Candida nappy rash (Infections and infestations) | 3 (3) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (2)
Conjunctivitis bacterial (Infections and infestations) | 4 (4) | 3 (4)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 3 (6) | 1 (2)
Gastroenteritis (Infections and infestations) | 3 (4) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 2 (3)
Hand-foot-and-mouth disease (Infections and infestations) | 4 (4) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 2 (2)
Otitis media (Infections and infestations) | 12 (17) | 3 (9)
Otitis media acute (Infections and infestations) | 9 (14) | 4 (10)
Otosalpingitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 7 (7) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 16 (39) | 7 (12)
Viral upper respiratory tract infection (Infections and infestations) | 9 (23) | 4 (12)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood lead increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Speech disorder developmental (Nervous system disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 3 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
Based on immunogenicity results from Part 1, Part 2 was not conducted. Results should be interpreted with caution due to the small sample size of Part 1 mRNA-1273.214 10 μg arm. Enrollment in Part 1 10 μg arm was halted as the target variant for the formulation was no longer a variant of concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT05584202/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT05584202/SAP_001.pdf